CLINICAL TRIAL: NCT07241481
Title: Comparing Two Different Attachments Retaining Mandibular Implant Overdenture Regarding Bone Changes and Occlusal Force Distribution (Randomized Clinical Trial)
Brief Title: Using Two Different Attachments (Equator Vs Ball and Sockets) Retaining Mandibular Implant Overdenture in Order to See Bone Changes and Occlusal Force Distribution
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Noha Taha Kamel Taha Alloush, Lecturer, Misr International University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 03410625
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Edentulous Alveolar Ridge In Mandible; Complete Edentulism; Dental Implant; Attachments; Implant Retained Overdenture; Edentulous Jaw
Keywords: Dental Implants; Attachments; Edentulous Ridge
MeSH Terms: conditions — Jaw, Edentulous

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ball & Socket Attachment (Active Comparator): On the 2nd stage, implants will be loaded with ball & socket attachments to retain overdenture
  Interventions: Procedure: Ball & Socket Attachment
- Equator Attachment (Experimental): On the 2nd stage, implants will be loaded with Equator attachments to retain overdenture
  Interventions: Procedure: Equator Attachment

INTERVENTIONS:
Procedure: Ball & Socket Attachment — Two implants will be restored using ball-and-socket attachment systems, with the mandibular denture retained over these attachments through corresponding metal housings
  Arms: Ball & Socket Attachment
Procedure: Equator Attachment — Two implants will be restored using Equator attachment systems, with the mandibular denture retained over these attachments through corresponding metal housings
  Arms: Equator Attachment

SUMMARY:
Alveolar ridge resorption is an unavoidable consequence in complete denture wearers due to limited retention and stability. Implant-retained overdentures enhance retention, stability, and masticatory performance while reducing ridge resorption and improving patients' quality of life.

Among attachment systems, ball-type anchors have long been favored for their simplicity and cost-effectiveness. However, the Equator attachment has emerged as a refined alternative, providing superior retention and stability for implant overdentures.

Functional performance can be evaluated through electromyography, which records masticatory muscle activity, and the T-Scan system, which analyzes occlusal force distribution and timing during dynamic occlusion. Additionally, bite force measurement serves as a key indicator of prosthetic efficiency and neuromuscular function, with implant-retained overdentures showing higher values than conventional dentures. This study aimed to compare bone level changes, occlusal force distribution in patients wearing mandibular implant overdentures retained by Equator and ball-and-socket attachments.

DETAILED DESCRIPTION:
All 24 patients will receive upper complete and lower complete overdentures. The upper complete denture will be mucosa supported while lower complete denture will be retained for by two dental implants in the inter-foraminal region. Patients will be divided into two equal groups; Group I will be retained by Ball and Socket attachment, while Group II will be retained by Equator attachment. Both groups will be functionally loaded after three months of insertion. This study aimed to compare bone level changes, occlusal force distribution in patients wearing mandibular implant overdentures retained by Equator and ball-and-socket attachments. Bone level changes will be measured using CBCT, While occlusal force will be measured using Tscan system.

ELIGIBILITY:
Inclusion Criteria:

* All patients age must range from 55- 60 years old.
* All patients' ridges should be covered with firm mucosa free from any signs of inflammation or ulceration and exhibit adequate height and width of the residual alveolar ridge.
* Patients should be free from any metabolic or bone disorder that contraindicate implant installation.
* All patients must have sufficient inter arch space

Exclusion Criteria:

1. Patients with oral or systemic diseases.
2. Patients with xerostomia or excessive salivation.
3. Patients with parafunctional habits (bruxism or clenching).
4. Heavy smoker or alcoholic patients.
5. Patients with history of temporo-mandibular dysfunction.
6. Patients with brain disorders or psychiatric disorders

Ages: 55 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Male patients aged between 55 and 60 years with completely edentulous maxillary and mandibular arches were included in the study. All participants demonstrated good oral hygiene, an Angle Class I maxilla-mandibular relationship, and adequate interarch space. The residual alveolar ridges were covered by firm, healthy mucosa without signs of inflammation, ulceration, or flabbiness.
Enrollment: 24 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-11-01 (Actual); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Marginal Bone Changes | it will be measured at denture insertion, 6 month, and 12 month later
  Marginal bone height changes around the two implants were evaluated through the software by measuring the distance from the alveolar crest to the implant apex in both coronal and sagittal views. The amount of bone loss was calculated by subtracting the measured distance between each radiographic evaluation made at the time of denture insertion and the recall appointments by superimposition of images and average was taken

SECONDARY OUTCOMES:
Occlusal force distribution measurement | it will be recorded at the time of prosthesis insertion, 6 months, and 12 months after denture insertion.
  Occlusal force distribution was done using the T-Scan™ Novus™, which consists of a sensor registering occlusal contacts, a data transferring module linked to a computer, and a software program to send data to the computer and visualize them on the monitor

CONTACTS AND LOCATIONS:
Locations (1):
- Oral and Dental Research Institute, National Research Center, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Study Protocol and Clinical Study Report
Supporting Information: Study Protocol, CSR
Time Frame: Start Date: After publication End Date: 3 years
Access Criteria: After publication through the corresponding author